CLINICAL TRIAL: NCT02142556
Title: The Efficacy and Safety of Once-daily Quetiapine Extended Release in Patients With Schizophrenia Switched From Other Antipsychotics
Brief Title: The Efficacy and Safety of Quetiapine XR in Patients With Schizophrenia Switched From Other Antipsychotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Chin-Bin Yeh, Chief, Associate Professor, Department of Psychiatry, Tri-Service General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00046
Record Dates: First submitted 2014-05-12; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine XR (Experimental): Patients had schizophrenia and fulfilled the criteria including having a score of 4 (moderate) or greater on any of the 7 items of the Positive and Negative Syndrome Scale (PANSS) Positive Symptom Subscale and needed to switch from previous antipsychotics due to insufficient efficacy or insufficient tolerability (N=61). They will receive the intervention of administration of quetiapine XR.
  Interventions: Drug: Administration of quetiapine XR

INTERVENTIONS:
Drug: Administration of quetiapine XR — The treatment was initiated with a 7-day cross-titration period. Previous antipsychotic medication was maintained at the original dose from day 1 to day 3; then reduced to 50% of the original dose from day 4 to day 7 and discontinued on day 8. Meanwhile, the patients started quetiapine XR with daily dose at 300 mg on day 1, 600 mg on day 2 and up to 800 mg after day 2. From day 8 until the end of the study, the dose of quetiapine XR was adjusted within 400-800 mg per day, depending on the clinical response and tolerability of the patients.

SUMMARY:
Purpose To evaluate the efficacy and safety of once-daily quetiapine extended release (XR) in patients with schizophrenia switched from other antipsychotics which were suboptimal due to insufficient efficacy or insufficient tolerability.

Methods:

This was a 12-week, open-label study conducted in the Chinese population in Taiwan. Quetiapine XR was administrated at 300 mg on day 1, 600 mg on day 2 and up to 800 mg after day 2. From day 8 until the end of the study, the dose of quetiapine XR was adjusted within 400-800 mg per day, depending on the clinical response and tolerability of the patients.

ELIGIBILITY:
Inclusion Criteria:

* The participants who were aged from 20 to 65 years and met the diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM-IV-TR) were eligible for the recruitment to the clinical trial.
* They also fulfilled the criteria including having a score of 4 (moderate) or greater on any of the 7 items of the Positive and Negative Syndrome Scale (PANSS) Positive Symptom Subscale and needed to switch from previous antipsychotics due to insufficient efficacy or insufficient tolerability.

Exclusion Criteria:

* Any DSM-IV-TR Axis I disorder other than schizophrenia, except comorbid obsessive-compulsive disorder, anxiety disorder, eating disorders or impulse control disorders if they had been stable and had not been primary focus of treatment over the previous 6 months
* An imminent risk of suicide or a danger to self or others
* Pregnancy or lactation
* Intolerance or lack of response to quetiapine IR
* Use of cytochrome P450 3A4 inhibitors or inducers in the 14 days preceding enrolment
* Administration of a depot antipsychotic injection within one dosing interval before recruitment
* Unstable or inadequately treated medical illness as judged by the investigator.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessments | 12 weeks
  The variable of the primary endpoint was the change from baseline to Week 12 in PANSS total and subscale score.

SECONDARY OUTCOMES:
Safety Assessments | 12 weeks
  The occurrence and severity of adverse events (AEs) will be recorded throughout the study to assess the tolerability of quetiapine XR, including AEs spontaneously reported by the patients or observed by the staff.

OTHER OUTCOMES:
Other Safety Assessments-the measure is a composite for metabolic disturbance | 12 weeks
  The patient's vital signs and body weight will be measured at screening and every visit schedule (week 1, 2, 4, 8, 12). An electrocardiogram and laboratory measurements including hematology and glycosylated hemoglobin (HbA1c) will be performed at enrolment and week 12.
Another efficacy assessment-CGI-S | 12 weeks
  Another efficacy endpoint was the difference from baseline to the end of study in Clinical Global Impression-Severity (CGI-S) score in the participants.
other safety assessments-the measure is a composite for EPS | 12 weeks
  Other scales used to evaluate the extrapyramidal symptoms (EPS) associated with the previous antipsychotics or quetiapine XR were Abnormal Involuntary Movement Scale (AIMS), Barnes-Akathisia Rating scale (BARS) and Simpson-Angus Scale (SAS). The use of anticholinergic medications during the treatment period will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Bin Yeh, M.D., Ph.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

REFERENCES:
- [Derived] Pan PY, Lee MS, Yeh CB. The efficacy and safety of once-daily quetiapine extended release in patients with schizophrenia switched from other antipsychotics: an open-label study in Chinese population. BMC Psychiatry. 2015 Jan 22;15:1. doi: 10.1186/s12888-014-0378-5. PMID 25609320